CLINICAL TRIAL: NCT07182994
Title: Immobilization During Peripheral Venous Catheter Placement in Paediatric Emergency Care: a Randomized Clinical Trial
Brief Title: Immobilization During Peripheral Venous Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Ana Martínez Serrano, Principal investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Immobilization catheter
Record Dates: First submitted 2025-08-29; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pediatrics; Immobilization
Keywords: pediatrics; emergency medical services; immobilization; catheter; nurses, pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elbow joint immobilization (Experimental): Pediatric patients undergo cannulation of a peripheral venous line with immobilization of the elbow joint
  Interventions: Procedure: Elbow joint immobilization
- arm restraint without immobilization of the elbow joint (Active Comparator): Pediatric patients undergo cannulation of a peripheral venous line with arm restraint, but the elbow joint is not immobilized.
  Interventions: Procedure: Arm restraint without elbow immobilization

INTERVENTIONS:
Procedure: Elbow joint immobilization — Immobilization of the elbow joint during peripheral venous line cannulation in pediatric patients on the success of the technique
  Arms: elbow joint immobilization
Procedure: Arm restraint without elbow immobilization — Use of arm restraint without immobilization of the elbow joint during peripheral venous line cannulation in pediatric patients.
  Arms: arm restraint without immobilization of the elbow joint

SUMMARY:
Aim: To determine the most effective type of upper limb immobilization in the cannulation of a peripheral venous line in the pediatric emergency department.

Methods: Randomized clinical trial with 322 patients conducted in a tertiary pediatric emergency. The impact of two types of restraints (immobilization of the elbow joint versus arm restraint, without immobilization of the elbow joint) on the success of the technique was analyzed. Multivariate analysis was used to analyze the impact of other variables (weight, age, movements, pain) on the success of the technique.

DETAILED DESCRIPTION:
A study will be conducted in a Spanish tertiary hospital to assess the holding technique for peripheral venous catheterization in pediatric patients presenting to the pediatric emergency department. The nursing staff will be responsible for implementing the study protocol, data collection, and subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients at emergency department that need a peripheral venous line

Exclusion Criteria:

* Critically ill patient

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 322 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
success of peripheral venous line cannulation on the first attempt | From enrollment to the end of the procedure (15 minutes)
  Percentage of successful cannulations on the first attempt, as assessed by the registered nurse.

SECONDARY OUTCOMES:
Number of attempts required | From enrollment to the end of the procedure (15 minutes)
  Number of cannulation attempts until successful catheterization.
Time to successful catheterization | From start of procedure until catheter placement (≤15 minutes)
  Time in minutes from first attempt to successful catheter placement
Nurse's assessment of patient's pain | Immediately after procedure
  Pain assessed by the nurse using a validated age-appropriate pediatric pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small sample of pediatric patients in a single hospital. Sharing the data could compromise confidentiality despite de-identification, and the main outcomes will be disseminated through peer-reviewed publications and conference presentations.